CLINICAL TRIAL: NCT05361915
Title: A Phase 2 Study of AbiVERtinib in Combination With Abiraterone in Patients With Metastatic Castration Resistant Prostate Cancer (Maverick Trial)
Brief Title: Study to Assess Abivertinib in Combination With Abiraterone in Metastatic Castration Resistant Prostate Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sorrento Therapeutics filed for chapter 11 bankruptcy.
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABV-RPC-201
Record Dates: First submitted 2022-04-15; First posted 2022-05-05 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic
Keywords: metastatic prostate cancer; castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abivertinib; abiraterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abivertinib - Abiraterone-naive (Experimental): Abiraterone-naive: Abivertinib 200 mg by mouth twice daily with abiraterone 1000 mg by mouth daily.
  Interventions: Drug: Abivertinib; Drug: Abiraterone
- Abivertinib - Abiraterone-progressing (Experimental): Abiraterone-progressing: Abivertinib 200 mg by mouth twice daily with abiraterone 1000 mg by mouth daily.
  Interventions: Drug: Abivertinib; Drug: Abiraterone

INTERVENTIONS:
Drug: Abivertinib — Abivertinib is a small molecule inhibitor
  Other Names: STI-5656
Drug: Abiraterone — Hormone-based chemotherapy

SUMMARY:
This is a phase 2, multicenter, open-label study to evaluate the efficacy of abivertinib with abiraterone in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
This is a phase 2, multicenter, open-label study to evaluate the efficacy of abivertinib with abiraterone in patients with metastatic castration-resistant prostate cancer via assessment of 6-month radiographic progression-free survival. The study will include two cohorts, abiraterone-naive and abiraterone-progressing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Metastatic disease as identified by imaging
* Progressive mCRPC as defined by: 1) castrate levels of serum testosterone < 50 ng/dL and 2) progressive disease
* Continued primary androgen deprivation with LHRH analogue (agonist or antagonist) if subject has not undergone bilateral orchiectomy
* Germline testing for HSD3B1. Confirmation of positivity for the adrenal-permissive HSD3B1(1245C) allele (germline heterozygous or homozygous) will be done centrally
* For abiraterone-progressing cohort, abiraterone must be the most immediate preceding line of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ and marrow function

Exclusion Criteria:

* Significant small cell or neuroendocrine component or histology
* Prior enzalutamide, apalutamide, or darolutamide exposure for either hormone sensitive or CRPC. Prior abiraterone is prohibited for the abiraterone-naïve combination cohort
* Prior BTK inhibitor treatment
* Need for concurrent CYP3A inducers and inhibitors
* Any condition including the presence of laboratory abnormalities that places the patient at unacceptable risk if the patient was to participate in the study
* Corrected QT interval calculated by the Fridericia formula per electrocardiogram within 14 days before Cycle 1 Day 1
* Any uncontrolled active systemic infection including any infection requiring systemic IV treatment that was completed ≤ 7 days before Cycle 1 Day 1, including active infection with COVID-19, defined as 10 days from the end of COVID-19 symptoms
* Have human immunodeficiency virus (HIV) infection, human T-cell leukemia virus type 1 (HTLV1) infection, or hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or are at risk for HBV reactivation (at risk for HBV reactivation is defined as being HBs antigen positive, or anti-HBc-antibody positive), or are positive for HBV deoxyribonucleic acid (DNA). HCV ribonucleic acid (RNA) must be undetectable by laboratory test
* Imminent or established spinal cord compression based on clinical and/or imaging findings
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks prior to Cycle 1 Day 1
* Major surgery within 4 weeks before Cycle 1 Day 1. Minor surgeries within 10 days before Cycle 1 Day 1. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible
* Radiation therapy within 2 weeks before Cycle 1 Day
* Participation in another investigational trial and received treatment within 4 weeks before Cycle 1 Day 1
* Any other active malignancy at the time of first dose of study treatment or diagnosis of another malignancy within 2 years prior to Cycle 1 Day 1 that requires active treatment, except locally curable cancers
* Unable to swallow tablets/capsules whole

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
6-month radiographic progression-free survival | baseline through study completion at up to approximately 63 months
  6-month radiographic progression-free survival (rPFS) will be assessed as defined by percent of subjects alive and without progression by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for measurable disease and Prostate Cancer Working Group 3 (PCWG3) criteria for bone metastases.

SECONDARY OUTCOMES:
Overall Response Rate | baseline through study completion at up to approximately 63 months
  Overall Response Rate (ORR) will be defined by percent of subjects alive and without progression by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of response | baseline through study completion at up to approximately 63 months
  duration of response will be defined as the time from the first documented response in patients with measurable disease to the date of progression or death due to any cause.
Prostate-Specific Antigen (PSA) progression | baseline through study completion at up to approximately 63 months
  Change in PSA as compared to baseline as defined by Prostate Cancer Working Group 3 (PCWG3) criteria
Safety and tolerability | baseline through study completion at up to approximately 63 months
  Safety and tolerability of abivertinib with abiraterone using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria.
Time to occurrence of first skeletal event | baseline through study completion at up to approximately 63 months
  Time to occurrence of first symptomatic skeletal event will be defined as the time from enrollment to the first symptomatic skeletal event defined as use of external beam radiotherapy to relieve skeletal symptoms or the occurrence of new symptomatic pathological bone fractures (vertebral or non-vertebral) or the occurrence of spinal cord compression or a tumor related orthopedic surgical intervention.
Time to first subsequent anti-cancer therapy | baseline through study completion at up to approximately 63 months
  Time to first subsequent anti-cancer therapy will be defined as the time from treatment discontinuation for any reason to start of subsequent anti-cancer therapy or death.
6-month radiographic progression-free survival (rPFS) | baseline through study completion at up to approximately 63 months
  6-month radiographic progression-free survival (rPFS) will be defined as the time from enrollment to progression by by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for measurable disease and and Prostate Cancer Working Group 3 (PCWG3) criteria for bone metastases or death, whichever occurs first.
Overall survival | baseline through study completion at up to approximately 63 months
  Overall survival will be defined as the time from enrollment to death

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (2):
- United States (2):
  - UCSD Moores Cancer Center, La Jolla, California
  - Cleveland Clinic, Cleveland, Ohio